CLINICAL TRIAL: NCT06900452
Title: A Randomized Controlled Trial to Investigate the Cognitive, Vascular, Neural and Biochemical Effects of Acute Pistachio Intervention in Older Adults
Brief Title: The Effect of Pistachio-Rich Breakfast Meals on Cognitive Function in Healthy Older Adults
Acronym: PACVAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-236-CW
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cognition
Keywords: Cognition; Pistachios; Vascular; Neural; Inflammation; Mood
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Macronutrient-matched placebo breakfast meal
  Interventions: Dietary Supplement: Placebo
- 0.5 servings of pistachio (Experimental): 0.5 servings of pistachio (15g) administered in breakfast meal
  Interventions: Dietary Supplement: 0.5 serving of pistachios
- 1 serving of pistachio (Experimental): 1 serving of pistachio (30g) administered in breakfast meal
  Interventions: Dietary Supplement: 1 serving of pistachios
- 2 servings of pistachio (Experimental): 2 servings of pistachio (60g) administered in breakfast meal
  Interventions: Dietary Supplement: 2 servings of pistachios

INTERVENTIONS:
Dietary Supplement: 0.5 serving of pistachios — The equivalent of 0.5 servings (15g) of shelled, roasted pistachio nuts, crushed and mixed into a muesli-based breakfast meal for consumption.
  Ingredients: 15g pistachio, 35g muesli base, 150g full fat natural yoghurt, 15g unsalted butter (melted), 10g unflavoured whey powder
  Arms: 0.5 servings of pistachio
Dietary Supplement: 1 serving of pistachios — The equivalent of 1 serving (30g) of shelled, roasted pistachio nuts, crushed and mixed into a muesli-based breakfast meal for consumption.
  Ingredients: 30g pistachio, 35g muesli base, 150g full fat natural yoghurt, 10g unsalted butter (melted), 5g unflavoured whey powder
  Arms: 1 serving of pistachio
Dietary Supplement: 2 servings of pistachios — The equivalent of 2 servings (60g) of shelled, roasted pistachio nuts, crushed and mixed into a muesli-based breakfast meal for consumption.
  Ingredients: 60g pistachios, 25g muesli base, 150g low fat natural yoghurt
  Arms: 2 servings of pistachio
Dietary Supplement: Placebo — Macronutrient-matched placebo breakfast meal. Ingredients: 40g muesli base, 150g full fat natural yoghurt, 25g unsalted butter (melted), 15g unflavoured whey powder
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of a breakfast meal containing varying serving sizes (doses) of pistachio nuts on cognitive function throughout the course of the day in healthy ageing adults aged 65-80.

DETAILED DESCRIPTION:
This crossover RCT investigates the acute postprandial effect (over a 6-hour period) of a breakfast meal containing varying serving sizes (doses) of pistachio nuts on the cognitive behaviour in healthy adults aged 65-80 years old. The study will also assess markers of inflammation and brain health by taking blood samples, and explore brain function (EEG) and blood flow (FMD) to understand how pistachio nuts may positively influence cognitive health. The study will involve a screening visit and four testing visits, with a week interval between each. On the evening prior to each test visit, participants are asked not to consume any food or drinks expect water, including tea/coffee and alcohol, after 8.30pm, and on the morning of test visits to only consume one slice of buttered white toast and a glass of water prior to attending the visit. During the four testing visits, cognitive and mood battery tests will be taken at baseline and then at 2-, 4- and 6-hour intervals following the consumption of the intervention meal. Blood draws are taken at the end of the day. For the subset of participants taking part in FMD, this will be measured at baseline, 2, 4 and 6 hours prior to cognitive testing. For those taking part in EEG, this data will be collected at 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* 65 - 80 years old
* Fruit & veg intake less than or equal to 4 servings per day
* Not regularly consuming more than 3 servings of fish per week
* Adequate English language and visual & auditory acuity to perform the cognitive tasks
* Normal BMI for age
* Normal MMSE performance between 26-30

Exclusion Criteria:

* Being diagnosed with psychological or psychiatric disorders
* ADHD or dyslexia
* Any food allergy or intolerance
* Use of medications and dietary supplements that may impact study results
* Antibiotic use within the last 3 months
* Adherence to vegan or vegetarian diets, or other specific diets that may impact study outcomes
* Being diagnosed with cardiometabolic disease (including type II diabetes and cardiovascular disease), or suffer from untreated hypertension or thrombosis related disorders
* Taking blood thinners

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Delayed recall (Rey Auditory Verbal Learning Task) | Baseline
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.
Delayed recall (Rey Auditory Verbal Learning Task) | 2 hours
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.
Delayed recall (Rey Auditory Verbal Learning Task) | 4 hours
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.
Delayed recall (Rey Auditory Verbal Learning Task) | 6 hours
  The RAVLT is a verbal learning task that presents participants with 15 words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. After 5 presentations, a new list (list B) is presented and recalled, and finally participants are asked (without hearing list A again) to recall as many words as they can from list A. After a 30 minute period, participants are asked to think back to the task and recall as many words as possible from list A only, providing a measure of delayed recall.

SECONDARY OUTCOMES:
Rate of learning (Rey Auditory Verbal Learning Task) | Baseline
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of learning (Rey Auditory Verbal Learning Task) | 2 hours
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of learning (Rey Auditory Verbal Learning Task) | 4 hours
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Rate of learning (Rey Auditory Verbal Learning Task) | 6 hours
  The RAVLT is a verbal learning task that presents participants with 15 sequential words (list A) 5 times, giving participants one minute after each presentation to recall as many words as they can from the list. Scores are recorded as a percentage of accuracy, and the rate of learning is determined through change in accuracy across the 5 recalls.
Word recognition (Rey Auditory Verbal Learning Task) | Baseline
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word recognition (Rey Auditory Verbal Learning Task) | 2 hours
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word recognition (Rey Auditory Verbal Learning Task) | 4 hours
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Word recognition (Rey Auditory Verbal Learning Task) | 6 hours
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Modified Attention Network Task (MANT) | Baseline
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Modified Attention Network Task (MANT) | 2 hours
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Modified Attention Network Task (MANT) | 4 hours
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Modified Attention Network Task (MANT) | 6 hours
  This task examines execution function, attention and inhibition. Participants respond to a centrally presented target arrow pointing to the left or the right by pressing the corresponding key on the keyboard. The target arrow is flanked by arrows that point in the same (congruent) or opposite (incongruent) direction. Previous studies have found that participants show larger latencies and more errors on incongruent trials when compared with congruent trials due to the conflicting interference of the incongruently facing arrows. Response latencies to congruent trials reflect processing speed, while errors on incongruent trials indicate susceptibility to interference. In this study participants will be presented with two blocks of the MANT - one normal block, and one block with the addition of serial 3s. In the serial 3s block, participants will be asked to count backwards in 3s out loud while continuing to perform the MANT, increasing the level of cognitive demand.
Task Switching Task | Baseline
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Task Switching Task | 2 hours
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Task Switching Task | 4 hours
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Task Switching Task | 6 hours
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii, 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Corsi Block Tapping Task | Baseline
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Corsi Block Tapping Task | 2 hours
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Corsi Block Tapping Task | 4 hours
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Corsi Block Tapping Task | 6 hours
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible by clicking with the mouse. Outcomes include number of correct sequences identified as a percentage of accuracy, and number of correct blocks identified (not necessarily in the correct sequence). Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
N-back task | Baseline
  The N-Back task is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. In this simplified 0-back version, participants respond when the target matches a fixed target specified at the beginning of the task (similar to a Go/No-Go task). Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG (6 hours only) in order to monitor change in brain activity in response to target trials. The N-Back was selected as it has been shown in previous work to elicit a strong P300 signal (see EEG as additional outcome).
N-back task | 2 hours
  The N-Back task is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. In this simplified 0-back version, participants respond when the target matches a fixed target specified at the beginning of the task (similar to a Go/No-Go task). Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG (6 hours only) in order to monitor change in brain activity in response to target trials. The N-Back was selected as it has been shown in previous work to elicit a strong P300 signal (see EEG as additional outcome).
N-back task | 4 hours
  The N-Back task is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. In this simplified 0-back version, participants respond when the target matches a fixed target specified at the beginning of the task (similar to a Go/No-Go task). Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG (6 hours only) in order to monitor change in brain activity in response to target trials. The N-Back was selected as it has been shown in previous work to elicit a strong P300 signal (see EEG as additional outcome).
N-back task | 6 hours
  The N-Back task is a measure of working memory where participants are instructed to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously. In this simplified 0-back version, participants respond when the target matches a fixed target specified at the beginning of the task (similar to a Go/No-Go task). Data will be analysed for both accuracy and reaction time on correct trials. For a subset of participants, this task will be conducted while recording EEG (6 hours only) in order to monitor change in brain activity in response to target trials. The N-Back was selected as it has been shown in previous work to elicit a strong P300 signal (see EEG as additional outcome).
EEG (ERPs & PSD) | 6 hours
  Event related potential (ERP) measure of P300 & N200 latency and amplitude will be assessed using EEG (electroencephalography) in a subset of participants during resting state (eyes open and closed) and during the N-Back task. Additionally, power for Alpha, Beta, Gamma, Delta, and Theta bands during performance of the N-Back task will be assessed in these participants.
  EEG data will be collected using Brain Products software and 16-channel active electrodes.
Blood markers | 6 hours
  Blood samples will be collected 6 hours post-intervention to measure to following serum markers: BDNF, irisin, IGF-1 and cytokines (IL-6, IL-10 and TNF-α). Samples will be analysed using enzyme-linked immunosorbent assays.
Flow mediated dilation (FMD) | Baseline
  A subset of participants will complete FMD assessment prior to each cognitive task battery (baseline, 2, 4 and 6 hours). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Flow mediated dilation (FMD) | 2 hours
  A subset of participants will complete FMD assessment prior to each cognitive task battery (baseline, 2, 4 and 6 hours). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Flow mediated dilation (FMD) | 4 hours
  A subset of participants will complete FMD assessment prior to each cognitive task battery (baseline, 2, 4 and 6 hours). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Flow mediated dilation (FMD) | 6 hours
  A subset of participants will complete FMD assessment prior to each cognitive task battery (baseline, 2, 4 and 6 hours). FMD is a non-invasive ultrasound technique that measures how the brachial artery dilates in response to increased blood flow following occlusion. Participants are required to lie down for 15 minutes before scanning commences. The procedure then takes 9 minutes: the brachial artery is first scanned for 1 minute, a blood pressure cuff is then inflated on the forearm for 5 minutes, before being released and the artery scanned for a further 3 minutes. This data will be analysed using Cardiovascular Suit. During FMD, laser doppler flowometry (LDF) will also be measured using the index finger of the right arm and analysed for % PORH (post occlusive reactive hyperaemia), measured in flux units .
Raven's Progressive Matrices | Baseline
  The Raven's is a non-verbal intelligence test designed to assess abstract reasoning and fluid intelligence which provides a single score (the sum of correct answers). Ravens will be included in the present study at baseline as a measure of IQ, which may later be utilised as a covariate when analysing the cognitive data.
Epic-Norfolk Food Frequency Questionnaire | Baseline
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
Blood pressure | Baseline
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Blood pressure | 2 hours
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Blood pressure | 4 hours
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.
Blood pressure | 6 hours
  Average (triplicate) resting brachial left arm cuffed systolic and diastolic blood pressure mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, PhD, Principal Investigator — University of Reading
Locations (1):
- Nutrition, Cognition & Health Lab, School of Psychology and Clinical Language Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All relevant study outcomes described in the Ethics Review Application Form, including demographics, anthropometrics, cognitive performance, blood tests FMD and EEG data, will be preserved and made available via a data repository, such as the University of Reading data repository, in anonymised form, so that they can be consulted and re-used by others.